CLINICAL TRIAL: NCT04858477
Title: Use of the Napoleon to Improve Polyp Measurement in Gastroenterology Fellows
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-01268
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Colonoscopy Patients + their Gastroenterology Fellows (Other): Inpatient and outpatient colonoscopies performed by fellows at NYU Langone Health, NYU Langone Hospital Brooklyn, Bellevue Hospital Center, and Manhattan VA Medical Center from October 2020 - March 2021. These will include all colonoscopies with polyps done in adults age 45 and above.
  Interventions: Other: Visual estimation of polyp size; Device: Napoleon measurement of polyp size

INTERVENTIONS:
Other: Visual estimation of polyp size — For each colonoscopy, a fellow will first visually estimate the polyp size
Device: Napoleon measurement of polyp size — For each colonoscopy, a fellow will first visually estimate the polyp size and then measure the polyp with Napoleon. The Micro-Tech Endoscopic Polyp Measurement Device named Napoleon is a small catheter with a 15mm ruler calibrated at 1mm intervals with 5mm demarcations. It is classified as a Class 1, 510(k) exempt device by the FDA.

SUMMARY:
This is a clinical trial assessing gastroenterology fellows' accuracy of colonic polyp measurement using a Micro-Tech Endoscopic Polyp Measurement Device named Napoleon. The study will evaluate the feasibility of Napoleon as a polyp measurement device. Investigators will collect data on inpatient and outpatient colonoscopies performed by fellows at NYU Langone Health, NYU Langone Hospital Brooklyn, Bellevue Hospital Center, and Manhattan VA Medical Center from May 2021 - May 2022 for 150 patients. Investigators will include all colonoscopies with polyps done in adults age 45 and above. For each colonoscopy, a fellow will first visually estimate the polyp size and then measure the polyp with Napoleon. Investigators will calculate the difference in polyp measurement between visual assessment and using Napoleon for each fellow year and compare differences among fellow years. Investigators will evaluate for changes in fellows' accuracy of polyp measurement with subsequent uses of Napoleon. Investigators will determine the proportion of cases with a change in the recommended surveillance interval based on polyp size. A survey will be given to all fellows to assess the level of ease with using Napoleon.

ELIGIBILITY:
Patients:

Inclusion Criteria:

1. Adult age 45 and above
2. Undergoing a colonoscopy performed by a gastroenterology fellow
3. Willingness and ability to provide informed consent

Exclusion Criteria:

1. History of not tolerating prior colonoscopies well or difficult colonoscopies (e.g. high sedative requirement)
2. Undergoing a diagnostic colonoscopy for inflammatory bowel disease or other known inflammatory/infectious process

An individual who meets any of the following criteria during the colonoscopy will be excluded from participation in this study:

1. Colonoscopy without polyps
2. Polyps not removed in entirety
3. Polyps with indeterminate size

An individual who meets any of the following criteria after the colonoscopy will be excluded from participation in this study:

1. Hyperplastic or non-adenomatous polyps on pathology report

Fellows

Inclusion Criteria:

1. NYU gastroenterology fellow
2. Willingness and ability to provide informed consent

Exclusion Criteria:

1. Not deemed to be medically trained and ready to perform a colonoscopy by supervising gastroenterology attending

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Difference in polyp measurement between visual assessment and using Napoleon in fellows | 6 months
Difference in accuracy of polyp measurement among fellow years | 6 months
Difference in fellows' accuracy of polyp measurement with subsequent uses of Napoleon | 6 months
Difference in polyp measurement between histology and using Napoleon | 6 months
Proportion of cases with a difference in the recommended surveillance interval based on polyp size | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Renee Williams, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - NYU Langone Hospital Brooklyn, Brooklyn, New York
  - Bellevue Hospital Center, New York, New York
  - Manhattan VA Medical Center, New York, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Renee.Williams@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: Requests may be directed to: Renee.Williams@nyulangone.org